CLINICAL TRIAL: NCT03549624
Title: Standardized Perioperative Management of Patients Operated With Acute Abdominal Surgery in a High-risk Emergency Setting
Acronym: SMASH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: NU-Hospital Organization, Sweden (Other)
Responsible Party: Principal Investigator, Mattias Prytz, MD, PhD. Head of Deperatment for Colorectal surgery, Department of Surgery, NU-Hospital Organization, Sahlgrenska University Hospital
Other Study IDs: Acute laparotomy NU
Record Dates: First submitted 2018-03-01; First posted 2018-06-08 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Laparotomy; Peritonitis; Ileus; Perforated Bowel; Acute Abdomen
MeSH Terms: conditions — Peritonitis; Ileus; Intestinal Perforation; Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: All adult (>18y) patients with the need of an acute laparotomy (within 6 hours) at NÄL.
  Patients will be treated with an perioperative regime/protocol consisting of:
  1. Early so called NEWS-monitoring (measuring of standard physiological parameters);
  2. Early start of antibiotics;
  3. Rapid (within 6 hours) start of operation;
  4. Goal-directed fluid therapy;
  5. Intensified post-operative monitoring;
  6. The presence of both surgical and anesthesiological specialists in the early care of the patients.
  Interventions: Other: Standardised protocol for the perioperative management in patients in need of an acute laparotomy
- Control group: All patients operated with an acute laparotomy at NÄL the years prior to the study will be retrospectively collected using the hospitals operation management database (Orbit©). Medical data will be collected from the patients' medical charts and outcome data (i.e. mortality, length of hospital stay, surgical complications, ICU-management etc.) will be registered

INTERVENTIONS:
Other: Standardised protocol for the perioperative management in patients in need of an acute laparotomy — A standardised protocol for the perioperative management of patients including early start of antibiotics and swift surgical intervention as well as an emphasis on repeated monitoring of physiological parameters pre- and post-operatively.
  Groups: Intervention group

SUMMARY:
The objective of the study is to handle patients with the need for an acute laparotomy according to a standardised perioperative protocol and to document the measurement as they are performed (i.e. adherence to the protocol) and to measure the outcome with regard to both short- (30 days) and long-term (3 and 12 months) mortality. Several secondary endpoints will be measured, such as: hospital stay, length of stay at an Intensive Care Unit (ICU), readmission to ICU and surgical complications according to the Clavien-Dindo score. These results will then be compared to published rates of mortality from the literature and to similar outcomes for a cohort of all patients operated at NÄL on the same indication the years prior to the project/study.

DETAILED DESCRIPTION:
200-250 acute laparotomies are performed annually at NÄL. The operations are performed for a number of reasons, where operation due to ileus; with- or without bowel strangulation; operation for acute peritonitis due to different kinds of stomach- or bowel perforation and re-operations for complications to elective surgery are the most common. A common trait for all these patients is that they are all susceptible to negative effect on organ functions on virtually all organ systems due to the underlying condition/disease for which they are being operated. This impact on organ functions include negative effects on circulation (cardiovascular system), respiration, renal function, hepatic function, coagulation and central nervous system. Sepsis is common and causes/contributes to the impaired organ functions. Multi Organ Failure (MOF) is sometimes present both pre- and postoperatively. Hence these patients are critically ill, and the outcome with regard to morbidity is severe and mortality rates are high with numbers between 14% to 90% in different populations with different age and comorbidity.

Standard care for these patients in a Swedish setting is a rapid anesthesiological assessment of the patient, preoperative resuscitation - if deemed necessary - followed by surgical intervention. Postoperative care and monitoring dependent on local facilities/routines and individual assessment of the patient and the patients postoperative needs by the surgeon and anaesthetist together.

Recent studies from the United Kingdom indicate that at more standardised protocol with emphasis on six different measures have the possibility to improve postoperative outcome with regard to short term (30 days) mortality. The measures at hand are not new nor untried but the combination of measures including the shortened time to surgery are shown to be beneficial for the patients. The measures are: 1. early so called NEWS-monitoring (measuring of standard physiological parameters); 2. Early start of antibiotics; 3. Rapid (within 6 hours) start of operation; 4. Goal-directed fluid therapy; 5. Intensified post-operative monitoring; 6. The presence of both surgical and anesthesiological specialists in the early care of the patients.

This kind of standardised perioperative protocols has not yet been implemented in Swedish health-care.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the need of an acute laparotomy at NÄL

Exclusion Criteria:

* Laparotomy planned in advance and without suspicion of an acute intraabdominal pathology.
* Abdominal wall hernias (with no suspicion of ileus or bowel ischemia)
* Appendectomy (Laparoskopically or open)
* Cholecystectomi (Laparoskopically or open)
* Acute thoracotomy
* Akute aortic surgery
* Planned second look-surgery (including change of open abdominal drapings/VAC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at the department of surgery at NÄL, with the need for an acute laparotomy.
Sampling Method: Probability Sample
Enrollment: 1435 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-06 (Estimated)

PRIMARY OUTCOMES:
Short term mortality | 30 days
  30 days overall mortality following acute laparotomy

SECONDARY OUTCOMES:
Long term mortality | 3 months
  3-months overall mortality following acute laparotomy
Long term mortality | 12 months
  12 months overall mortality following acute laparotomy
Hospital stay | 12 months
  Length of hospital stay for survivors following acute laparotomy
Intesive care need | 12 months
  The need for ICU-care following acute laparotomy
Intesive care need | 12 months
  The need for readmission to the ICU following acute laparotomy
Surgical complications | 12 months
  Surgical complications (according to the Clavien-Dindo score) following acute laparotomy

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Prytz, MD, PhD, Principal Investigator — Sahlgrenska University Hospital an NU Hospital Oranization
Locations (1):
- Department of Surgery, NU-Hospital/NÄL, Trollhättan, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tengberg LT, Bay-Nielsen M, Bisgaard T, Cihoric M, Lauritsen ML, Foss NB; AHA study group. Multidisciplinary perioperative protocol in patients undergoing acute high-risk abdominal surgery. Br J Surg. 2017 Mar;104(4):463-471. doi: 10.1002/bjs.10427. Epub 2017 Jan 23. PMID 28112798
- [Result] Huddart S, Peden CJ, Swart M, McCormick B, Dickinson M, Mohammed MA, Quiney N; ELPQuiC Collaborator Group; ELPQuiC Collaborator Group. Use of a pathway quality improvement care bundle to reduce mortality after emergency laparotomy. Br J Surg. 2015 Jan;102(1):57-66. doi: 10.1002/bjs.9658. Epub 2014 Nov 10. PMID 25384994
- [Derived] Jansson Timan T, Hagberg G, Sernert N, Karlsson O, Prytz M. Mortality following emergency laparotomy: a Swedish cohort study. BMC Surg. 2021 Aug 11;21(1):322. doi: 10.1186/s12893-021-01319-8. PMID 34380437